CLINICAL TRIAL: NCT02289976
Title: Talar Avascular Necrosis: Surgical Angiogenesis Compared to Core Decompression With Osseous Autografting
Brief Title: Talar Avascular Necrosis: Surgical Angiogenesis vs. Core Decompression
Acronym: TalarAVN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BG Trauma Center Ludwigshafen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BGU-01/14
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Avascular Necrosis of Bone
Keywords: talar avascular necrosis; osteochondrosis dissecans; femoral condyle
MeSH Terms: conditions — Osteonecrosis; Osteochondritis Dissecans

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- femoral condyle (Active Comparator): Core decompression of the talar avascular necrosis followed by free microvascular femoral condyle grafting
  Interventions: Procedure: core decompression
- core decompression (Active Comparator): Core decompression and nonvascularized autograft from the iliac crest
  Interventions: Procedure: core decompression

INTERVENTIONS:
Procedure: core decompression — Drilling of the avascular necrosis of the talus by 10mm drill under x-ray control

SUMMARY:
The purpose of this study is to determine if surgical angiogenesis performed in talar avascular necrosis by free microvascular bone grafts from the medial femoral condyle is a superior technique compared to core decompression and nonvascularized osseous autografts.

DETAILED DESCRIPTION:
The aim of this prospective randomized clinical trial is the comparison of two surgical treatment options for talar avascular necrosis (analogical to Ficat and Arlet stage II and III). The randomized study design allows direct comparability of the outcome after either core decompression and nonvascularized osseous autografting from the iliac crest or core decompression and osseous autografting with a free microvascular medial femoral condyle.

Talar avascular necrosis is caused by osseous malperfusion leading to malnutrition and destruction of the talar bone. The extend of this malperfusion is variable and can be categorized in 4 stages. The osseous defects can remain without consequences (stage I) or lead to irreversible talar destruction. The current treatment option for stage II and III is the core decompression followed by osseous auto grafting from the iliac crest. Reducing the intraosseal pressure and filling the drill holes with the nonvascularized bone graft can lead to reperfusion of the talus.

A new technique is to fill the drill hole with a vascularized bone graft from the medial femoral condyle, using microvascular anastomosis. This procedure has already been approved for the treatment of avascular necrosis and malperfusion of the carpus (lunate and scaphoid) as well as the femoral head.

Patients are examined preoperative as well as 3, 6 and 12 month after operation, documenting the active range of motion and pain sensation while resting and on activity. Well established scores like the AOFAS Ankle-Hindfoot Score and the Lower Extremity Functional Scale are used to get subjective and objective informations about patients' daily life and postoperative satisfaction. X-Rays are taken at the same stages. MRIs of the ankle joint with contrast agent are performed before as well as 6 and 12 months after surgery.

Statistical analysis is performed using the Statistical Package for the Social Sciences (SPSS). The Study protocol has been approved by the Ethics Commission of Rheinland-Pfalz. Interventions are done according to the declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* patients with talar avascular necrosis without response to non-surgical treatment (immobilization) and with need for surgical intervention (Ficat and Arlet stage II and III; Berndt and Harty stage II and III)

Exclusion Criteria:

* talar avascular necrosis stage I (without need for surgical intervention)
* surgical revascularization in the past
* participation in a different study
* pregnancy
* peripheral artery occlusive disease
* drug associated talar avascular necrosis
* ongoing steroid therapy or chemo therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Pain reduction | pre operation; 3, 6, 12 months post operation
  measured by visual anloge scale

SECONDARY OUTCOMES:
Revascularization of the talus in the MRI | 6, 12 month post operation
  by ARCO-Criteria
Lower Extremity Functional Scale | pre operation; 3, 6, 12 month post operation
American Orthopaedic Foot and Ankle Society (AOFAS-) Ankle-Hindfoot-Score | pre operation; 3, 6, 12 month post operation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kremer, Phd, MD, Study Director — BG Trauma Center Ludwigshafen
Locations (1):
- BG Trauma Center Ludwigshafen, Ludwigshafen am Rhein, Rhineland-Palatinate, Germany

REFERENCES:
- [Background] Ficat RP. Idiopathic bone necrosis of the femoral head. Early diagnosis and treatment. J Bone Joint Surg Br. 1985 Jan;67(1):3-9. doi: 10.1302/0301-620X.67B1.3155745. No abstract available.
- [Background] BERNDT AL, HARTY M. Transchondral fractures (osteochondritis dissecans) of the talus. J Bone Joint Surg Am. 1959 Sep;41-A:988-1020. No abstract available. PMID 13849029
- [Result] Doi K, Sakai K. Vascularized periosteal bone graft from the supracondylar region of the femur. Microsurgery. 1994;15(5):305-15. doi: 10.1002/micr.1920150505. PMID 7934797
- [Result] Hussl H, Sailer R, Daniaux H, Pechlaner S. Revascularization of a partially necrotic talus with a vascularized bone graft from the iliac crest. Arch Orthop Trauma Surg. 1989;108(1):27-9. doi: 10.1007/BF00934153. PMID 2643938